CLINICAL TRIAL: NCT04199520
Title: Compare the Efficacy of Surgery Combined With Systemic Therapy and Pure Systemic Therapy in Patients With Stage Ⅳ Breast Cancer
Brief Title: Compare the Efficacy of Surgery Combined With Systemic Therapy and Pure Systemic Therapy in Breast Cancer Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: In clinical treatment, most patients with stage IV breast cancer received surgical treatment, which made it difficult to enroll this project, so this study was terminated.
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HNCH-BC003
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2019-12

CONDITIONS: Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgery combined with systemic therapy (Experimental): surgery combined with systemic therapy
  Interventions: Combination Product: surgery combined with systemic therapy
- systemic therapy (Active Comparator): systemic therapy
  Interventions: Other: systemic therapy

INTERVENTIONS:
Combination Product: surgery combined with systemic therapy — surgery combined with systemic therapy
  Arms: surgery combined with systemic therapy
Other: systemic therapy — systemic therapy
  Arms: systemic therapy

SUMMARY:
The purpose of this study is to compare the effect of primary resection combined with systemic therapy and pure systemic therapy on the overall survival of patients with stage Ⅳ breast cancer.

DETAILED DESCRIPTION:
In developing countries, the proportion of breast cancer patients who have a stage IV diagnosis at the first diagnosis can be as high as 25%. For advanced breast cancer, previous views have suggested that surgery as one of the palliative treatments does not improve patient survival. The proportion of patients undergoing surgery for stage IV breast cancer has gradually decreased over the past 30 years. At present, there is still no clear recommendation and guidance in common clinical guidelines for the primary surgery for stage IV breast cancer. Some retrospective studies suggest that surgery can improve the survival of advanced breast cancer, but the results of prospective studies are inconclusive, and surgery is still not a routine choice for stage IV breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* • Sign the informed consent

  * ages 18-70, female;
  * Breast cancer meets the following criteria:
* Histologically diagnosed invasive breast cancer, measure distant metastases with local standard assessment methods;
* Known hormone receptors and HER-2 status (ER, PR and HER2);

  * Eastern Cooperative Oncology Group (ECOG) performance status score ≤1;
  * Estimated patient survival beyond 1 year;
  * The time from diagnosis or systemic treatment to randomization does not exceed 1 year;
  * According to RECIST 1.1, patients receiving chemotherapy or endocrine therapy are effective, including complete remission, partial remission, or stabilization. If the patient only receives endocrine therapy, the time is not less than 6 months; when receiving chemotherapy, the number of cycles is not less than 4 cycles;
  * HER2-positive patients: the proportion of patients receiving targeted therapy is not less than 80% of the total HER2-positive patients;
  * Patients had no obvious surgical contraindications before randomization;
  * Researchers judge that they can comply with the research protocol

Exclusion Criteria:

* • Double breast cancer;

  * Progression of metastases after systemic treatment;
  * Poorly controlled brain metastases, liver metastases and multiple metastases;
  * History of local breast radiotherapy after diagnosis;
  * Have a history of other malignancies within 5 years prior to screening, with cervical cancer in situ treated properly except for non-melanoma skin cancer or stage I uterine cancer;
  * Have undergone a major breast cancer-free surgical procedure within 4 weeks before randomization, or the patient has not fully recovered from such a surgical procedure;
  * Have severe comorbidities or other comorbid conditions that interfere with planned treatment, or any other condition in which the investigator does not consider the patient suitable for participation in the study.
  * Patients can withdraw informed consent at any time;
  * pregnancy;
  * The sponsor has determined that a major protocol violation that could compromise patient safety;
  * Patients' non-compliance with protocol requirements on multiple occasions;
  * The investigator believes that withdrawal from the trial will be of greatest benefit to the patient.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
OS | up to 2 year
  The time from diagnosis to death

SECONDARY OUTCOMES:
PFS | up to 2 year
  The time from randomization to disease progression or death, including local PFS and distant PFS Local PFS refers to the time from randomization of patients to local or regional lymph node recurrence in the surgical group or local or regional lymph node progression in the non-surgical group. distant PFS refers to the time from randomization of a patient to local or distant distant disease progression or death.
BCSS (Breast Cancer Specific Survival) | up to 2 year
  The time from the random start of a patient to death due to breast cancer, excluding deaths caused by other causes

CONTACTS AND LOCATIONS:
Overall Officials: Jiujun Zhu, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China